CLINICAL TRIAL: NCT05985499
Title: A Randomized Parallel-controlled Study Comparing the Ileostomy "Dumpling Suture Method" With Traditional Suture Method in Rectal Anterior Resection Surgery With Specimen Extraction Via Stoma (NOSES With Specimen Extraction Via Stoma)
Brief Title: A Randomized Parallel-controlled Study Comparing the Ileostomy "Dumpling Suture Method" With Traditional Suture Method in Rectal Anterior Resection Surgery With Specimen Extraction Via Stoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tingyu Wu, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XHEC-C-2023-022-2
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-04

CONDITIONS: Ileostomy; Complications
Keywords: ileostomy; complications; NOSES; stoma suture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Dumpling suture" for ileostomy (Experimental): The stoma is fixed with sutures in a skin fold method, and the incision is progressively reduced in a process similar to the process of folding and pinching the Chinese small dumplings. This procedure may reduce stoma complications by progressively reducing the incision and realizing the effect of hiding the skin incision.
  Interventions: Procedure: Suturing of ileostomy using "Dumpling suture method"
- Traditional suture for ileostomy (Other): The stoma was fixed at the skin using traditional sutures. The incision is narrowed by 2-3 interrupted sutures at the distal and proximal ends of the skin incision on the abdominal wall. The stoma is then fixed at the right lower abdominal incision with sutures.
  Interventions: Procedure: Suturing of ileostomy using Traditional suture method

INTERVENTIONS:
Procedure: Suturing of ileostomy using "Dumpling suture method" — Suturing of ileostomy using "Dumpling suture method"
  Arms: "Dumpling suture" for ileostomy
Procedure: Suturing of ileostomy using Traditional suture method — Suturing of ileostomy using Traditional suture method
  Arms: Traditional suture for ileostomy

SUMMARY:
Natural Orifice Specimen Extraction Surgery (NOSES), which involves obtaining specimens from the abdominal cavity without any incisions, has attracted much attention in recent years, and it has been widely popularized in the treatment of rectal cancer because of its postoperative non-incision, advantages of less trauma, quicker recovery, and postoperative aesthetics. Anastomotic fistula is a serious complication of rectal cancer surgery. For patients at high risk of anastomotic fistula, prophylactic ileostomy is often performed intraoperatively to divert feces and protect the anastomosis. For such patients, rectal anterior resection surgery with specimen extraction via stoma (NOSES with specimen extraction via stoma) is usually performed, borrowing a prophylactic stoma incision to retrieve the specimen, and also realizing the absence of additional abdominal incision. However, this procedure is prone to stoma infection and has a high complication rate (20-40%), which limits the popularization of NOSES surgery and is an urgent clinical problem. Our center has proposed a new stoma closure method (Dumpling Suture Method), which reduces the size of the incision by folding the suture to achieve the effect of hiding the skin incision and reduce stoma infection. In our previous study, 17 cases of the new procedure were completed in our center, and 25 patients with stoma closure by the traditional method were included in the same period for control purposes. After six months of follow-up, we found that the "dumpling suture method" significantly reduced the incidence of stoma complications compared with the traditional suture method (5.8% vs. 36%), and no additional adverse effects were observed. This is a single-center, open-label, randomized, parallel-controlled clinical study. The primary endpoint is stoma complication rate within 30 days postoperatively. In this study, we aim to evaluate the efficacy and safety of the "dumpling suture method " compared with the traditional stoma suture in reducing postoperative stoma complications through a randomized parallel controlled clinical trial, which is of great significance for the improvement of the rectal NOSES procedure and the reduction of the incidence of stoma complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for rectal anterior resection surgery with specimen extraction via stoma
2. No serious systemic infection or immunosuppression
3. Patients aged above 18 years and below 100 years
4. Eastern Cooperative Oncology Group Performance Status: 0-1
5. Expected survival time > 6 months
6. Patient participate voluntarily and sign an informed consent form

Exclusion Criteria:

1. Patients who do not require a prophylactic stoma after preoperative evaluation
2. Any skin infectious disease of the abdominal wall
3. Surgery less than 1 month from the last chemotherapy
4. Previously underwent any other stoma surgery
5. Presence of a serious active or uncontrollable infection requiring systemic therapy
6. Previous history of definite neurological or psychiatric disorders
7. Patient may not be able to complete the study for other reasons, or who the investigator believes should not be included

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Complication rate of stoma | Within one month after surgery
  Observe and assess for stoma complications

SECONDARY OUTCOMES:
Stoma DET（Discoloration，Erosion and Tissue overgrowth） score | Within one month after surgery
  Measure the state of the skin around the stoma and the corresponding lesion area, ranging from 0-15, higher scores mean a worse outcome of stoma
Stoma Pain Score | Within one month after surgery
  Measurement of stoma pain level using numerical rating scale，ranging from 0-10, higher scores mean a worse outcome of pain
Quality of life scale score for patients with stoma | Day 30 after surgery
  Measurement of quality of life for patients with stoma using City of Hope Quality of Life-Ostomy Questionnaire (CHO-QOL-OQ), ranging from 0-3200, higher scores mean a worse outcome of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tingyu Wu, Doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
In this study personal information and data such as patient history, physical examination results, surgical records, and study questionnaire data will be collected. These data will be used to evaluate the efficacy and safety of the new procedure and for academic publication. The researcher will treat the patients' personal data confidentially and anonymize the data and information in any public release of the results of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR